CLINICAL TRIAL: NCT01351974
Title: Cohort Study of Axillary Recurrences and Survival After Negative Negative Sentinel Node Biopsy Without Completion Axillary Clearance
Brief Title: Sentinel Node Biopsy in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Swedish Cancer Society (Other)
Responsible Party: Leif Bergkvist, Centre for Clinical Research, Uppsala University
Other Study IDs: 00-053
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2000-06

CONDITIONS: Recurrence; Breast Cancer
Keywords: breast cancer; sentinel lymph node biopsy; axillary recurrence
MeSH Terms: conditions — Recurrence; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Routine specimens from the surgery are kept at the respective pathology departments
Oversight: Data Monitoring Committee: No

SUMMARY:
Axillary lymph node dissection (ALND) was previously the standard axillary staging procedure in breast cancer patients. However, ALND is accompanied by a considerable morbidity, and sentinel lymph node biopsy (SLNB) evolved as a mean to decrease this morbidity. Between September 2000 and January 2004 breast cancer patients were included in the Swedish Sentinel Node Multicenter Cohort Study with the intent of studying axillary recurrence after negative SLNB for patients in which completion ALND were omitted. The patients were followed prospectively and events (local, regional and distant recurrences and deaths) were registered. The primary endpoint was axillary recurrence and secondary endpoints were disease-free, cancer-specific and overall survival.

DETAILED DESCRIPTION:
Axillary lymph node dissection (ALND) was previously the standard axillary staging procedure in breast cancer patients. However, ALND is accompanied by a considerable morbidity, including seroma formation, lymphedema, neuropathy of the arm with numbness, stiffness, impaired shoulder movement and pain. Sentinel lymph node biopsy (SLNB) has evolved as a mean to decrease this morbidity, and validation studies have demonstrated the accuracy of the method.

With the intent of studying axillary recurrence after negative SLNB for patients in which completion ALND were omitted, consecutive breast cancer patients were included in the Swedish Sentinel Node Multicenter Cohort Study between September 2000 and January 2004.

Patients with a unifocal, invasive breast cancer less than 3 cm in diameter were eligible for enrollment. Exclusion criteria were palpable regional lymph nodes, neoadjuvant chemo- or radiotherapy, pregnancy, known allergic reactions to blue dye or isotope, previous surgery in the ipsilateral breast, and preoperatively diagnosed tumor multifocality.

Surgical procedure:

After the preoperative injection of 40-60 mBq Technetium-99 nanocolloid (Solco Nanocoll®) and 1 ml blue dye (Patent Blue V®), sentinel lymph node (SLN) biopsy was performed. If no sentinel node could be identified, ALND of levels I and II was performed. A completion ALND was also performed in the event of a positive SLN biopsy, if lymph nodes clearly suspicious of metastasis were detected during surgery, or if the primary tumor in the breast was found to be multifocal on pathological examination.

Pathological assessment:

Frozen sections were obtained from each SLN and examined peroperatively. If a sentinel lymph node was smaller than 4 mm, two sections were analyzed separately. Nodes larger than 4 mm were bisected, and two sections from each half analyzed. According to the study protocol, at least three sections were prepared from the sentinel node or each part of a bisected node for definitive histopathology. Sections were stained with haematoxylin and eosin (HE). If no cancer cells were detected, immunohistochemistry (IHC) with cytokeratin antibodies was also performed.

Non-sentinel lymph nodes were examined by routine staining (HE) according to the protocol of each pathology department.

Treatment and follow-up:

Adjuvant treatment combinations were given according to national and regional treatment guidelines, based on tumor characteristics, lymph node status, and surgical treatment. Patients with isolated tumor cells were regarded as lymph node-negative. If breast-conserving surgery had been performed, radiation therapy to the breast was given, which was extended to include the regional lymph nodes in case of axillary lymph node metastases.

Chemotherapy was offered to all patients with lymph node metastases or those with a combination of unfavorable primary tumor characteristics (large tumor, high Elston score, progesterone receptor negativity), after consideration of their general health. Endocrine therapy was offered to all patients with estrogen or progesterone receptor-positive tumors larger than 10 mm. The actual reported adjuvant treatment is controlled for in the analyses.

Patients were followed prospectively. The research protocol postulated an annual follow-up with mammography and clinical examination.

After enrollment, data sheets, including information on primary tumor characteristics, number of sentinel and non-sentinel lymph nodes with and without metastasis, and given adjuvant treatment, were computerized. The study was approved by the ethics committee of Karolinska Institutet, Stockholm, and each region's local ethics committee. All patients gave written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Primary invasive breast cancer

Exclusion Criteria:

* Preoperatively diagnosed axillary metastases
* Multifocal tumors
* Tumors > 3 cm
* Impalpable tumors
* Earlier resection of the tumor
* Neoadjuvant treatment
* Pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with primary breast cancer in Swedish hospitals
Sampling Method: Non-Probability Sample
Enrollment: 3369 (Actual)
Dates: Start 2000-09; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Axillary recurrence after negative sentinel node biopsy | 5 years
  Prospective follow-up of axillary recurrences in patients with negative sentinel lymph node biopsy in which completion axillary lymph node dissection were omitted

SECONDARY OUTCOMES:
Survival | 5 years
  Survival (disease-free, cancer-specific and overall) in the sentinel lymph node biopsy cohort

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bergkvist, M.D. Ph.D., Principal Investigator — Centre for Clinical Research, Uppsala University
Locations (1):
- Centre for Clinical Research, Uppsala University, Västerås, Sweden

REFERENCES:
- [Result] Andersson Y, Frisell J, Sylvan M, de Boniface J, Bergkvist L. Breast cancer survival in relation to the metastatic tumor burden in axillary lymph nodes. J Clin Oncol. 2010 Jun 10;28(17):2868-73. doi: 10.1200/JCO.2009.24.5001. Epub 2010 May 10. PMID 20458033
- [Result] Bergkvist L, de Boniface J, Jonsson PE, Ingvar C, Liljegren G, Frisell J; Swedish Society of Breast Surgeons. Axillary recurrence rate after negative sentinel node biopsy in breast cancer: three-year follow-up of the Swedish Multicenter Cohort Study. Ann Surg. 2008 Jan;247(1):150-6. doi: 10.1097/SLA.0b013e318153ff40. PMID 18156935